CLINICAL TRIAL: NCT00368030
Title: Depression Response to Eszopiclone in Adults With Major Depressive Disorder (DREAMDD): A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 8-Week, Safety & Efficacy Study of Eszopiclone 3 mg Compared to Placebo in Subjects With Insomnia Related to MDD Acronym: DREAMDD
Brief Title: A Study of Eszopiclone in Subjects With Insomnia Related to Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190-052
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Insomnia; Depressive Disorder, Major
Keywords: Insomnia related to major depressive disorder.
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depressive Disorder, Major | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Eszopiclone 3 mg QD
  Interventions: Drug: Eszopiclone
- B (Placebo Comparator): Placebo tablet
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone 3 mg QD
  Other Names: Lunesta, (S)-Zopliclone
  Arms: A
Other: Placebo — Placebo tablet
  Arms: B

SUMMARY:
The purpose of this study is to evaluate subjective sleep efficacy in subjects with insomnia related to major depressive disorder.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled, parallel group study. The study consists of two groups of subjects with major depression treated for ten weeks with a common antidepressant regimen, 20-40 mg of fluoxetine hydrochloride per day; and randomized to receive (in addition) either eszopiclone 3 mg or placebo for eight weeks. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject must understand the purpose of the study and be willing to adhere to the study schedule and procedures described in this protocol.
* Subject must be 21 to 64 years of age (inclusive) on the day of signing consent.
* Subject must meet criteria for a primary and principal diagnosis of Major Depressive Disorder.
* Subject's current depressive episode is at least 2 weeks but not longer than 6 months in duration.
* Subject must meet criteria for insomnia related to MDD and the symptoms of insomnia must not pre-date the symptoms of MDD by more than 10 weeks.
* Subject must report a sleep onset time of > 30 minutes, and wake time after sleep onset of > 45 minutes, and < 6.5 hours of total sleep time at least three times a week over the previous month.
* Subject must take the Hamilton-D-17 scale and have a protocol pre-specified minimum score.
* Subject must have no known clinically significant abnormal laboratory, ECG, or physical examination findings at screening.
* Subject must meet one of the following conditions:
* Subject is not taking antidepressant medications at the time of study start.
* Subject is taking a sub-therapeutic dose of antidepressant or other disallowed psychotropic medication and with the approval of the investigator agrees to taper off of this medication, prior to completion of screening assessments at study start.

Exclusion Criteria:

* Female subject is pregnant, lactating or within 6 months post partum.
* Subject has known sensitivity to any selective SSRI, zopiclone, or eszopiclone.
* Subject has history of major depressive disorder that was refractory to treatment with SSRIs.
* Subject has a current primary psychiatric diagnosis of any of the following disorders: dementia, delirium, schizophrenia, psychosis, other psychotic disorders, dysthymic disorder; bipolar disorders; cyclothymic disorder, other mood disorders, nocturnal panic disorder, primary anxiety disorders, primary panic disorders or any other psychiatric disorder that would compromise the investigator's ability to evaluate the safety and efficacy of the study medication.
* Note: Subjects with Sexual and Gender Identity Disorders or other non-psychotic disorders will be considered on a case-by-case basis. Subjects with MDD and a secondary diagnosis of generalized anxiety disorder, panic disorders other than nocturnal panic disorder or seasonal affective disorder will be allowed.
* Subject has any of the following Personality Disorders diagnoses: schizotypal, schizoid, borderline personality disorder; mental retardation or any other personality disorder that would compromise the investigator's ability to evaluate the safety and efficacy of the study medication.
* Subject has difficulties in sleep initiation or maintenance associated with known medical diagnosis [e.g. sleep apnea, restless leg syndrome (RLS), or periodic leg movement syndrome (PLMS)], or has any condition that has or may affect sleep [(e.g., chronic pain, benign prostatic hypertrophy (BPH)].
* Subject has any clinically significant unstable medical or neurologic abnormality, unstable chronic disease, or a history of a clinically significant abnormality of the cardiovascular, respiratory, hepatic, or renal systems.
* Subject has a disorder or history of a condition (e.g., malabsorption, gastrointestinal surgery) that may interfere with drug absorption, distribution, metabolism, or excretion.
* Subject has a history of malignancy within 5 years, or current malignancy, except for non-melanoma skin cancer.
* Subject has a history of drug or alcohol abuse or dependence in the past 6 months or positive urine drug and alcohol test at screening.
* Subject is participating in, has participated in, or plans to participate in any investigational drug study within 30 days prior to screening until the end of this study.
* Subject has history of circadian rhythm disorder, or travels across >3 time zones on a regular basis.
* Subject is known to be seropositive for Human Immunodeficiency Virus (HIV).
* Subject has used any drugs known or suspected to affect hepatic or renal clearance capacity within a period of 30 days prior to screening.
* Subject is unwilling to refrain from drinking alcoholic beverages during study participation.
* Subject is a rotating or third/night shift worker.
* Subject is a staff member or relative of a staff member.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 545 (Actual)
Dates: Start 2004-01; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Mean subjective wake time after sleep onset (WASO) | 1 week

SECONDARY OUTCOMES:
Time to onset of 30% antidepressant response using the HAM-D-6 (Bech)
Mean WASO | Weeks 2, 3, 4, 6 and 8
Mean subjective total sleep time (TST) | Weeks 1, 2, 3, 4, 6, and 8
Mean subjective sleep latency (SL) | Weeks 1, 2, 3, 4, 6, and 8
Mean number of awakenings | Weeks 1, 2, 3, 4, 6, and 8
Quality and depth of sleep | Weeks 1, 2, 3, 4, 6 and 8
Daytime alertness | Weeks 1, 2, 3, 4, 6 and 8
Ability to concentrate | Weeks 1, 2, 3, 4, 6 and 8
Physical well-being | Weeks 1, 2, 3, 4, 6 and 8
Ability to function | Weeks 1, 2, 3, 4, 6, and 8
average rebound and withdrawal effects will be analyzed for each of the subjective sleep endpoints | Weeks 1, 2, 3, 4, 6, and 8
Time to onset of 50% antidepressant response using the HAM-D-6 (Bech) | Weeks 1, 2, 3, 4, 6, and 8
Time to onset of 50% and 30% antidepressant responses using the HAM-D-6 (Maier) | Weeks 1, 2, 3, 4, 6, and 8
Change in the HAM-D-6 (Bech) and HAM-D-6 (Maier) from baseline to each visit | Weeks 1, 2, 3, 4, 6, and 8
Change in the HAM-D-17 from baseline | Weeks 4 and 8
Symptom Questionnaire (SQ) Score (Depression Subscale) | Weeks 1, 2, 3, 4, 6, and 8
Daily Telephone Assessment (DTA) Score | Weeks 1, 2, 3, 4, 6, and 8
Change in HAM-D-6 (Bech), HAM-D-6 (Maier), HAM-D-17, SQ, and DTA during the wash-out phase until end of study | Weeks 8 and 10
SF-36 Score | Weeks 4, 8, and 10
Work Limitations Questionnaire (WLQ) Score | Weeks 2, 4, 8, and 10
Epworth Sleepiness Scale (ESS) | Weeks 1, 2, 3, 4, 6, 8, and 10
Insomnia Severity Index (ISI) score | Weeks 2, 4, 8, and 10
Clinical Global Impression | Weeks 1, 2, 3, 4, 6, 8, and 10
Safety will be assessed by physical examinations, a standard 12-lead ECG, vital signs, clinical laboratory assessments and AE reporting | Weeks 1 through 10

CONTACTS AND LOCATIONS:
Locations (65):
- United States (65):
  - Birmingham, Alabama
  - Peoria, Arizona
  - Tucson, Arizona
  - Fayetteville, Arkansas
  - Garden Grove, California
  - Irvine, California
  - Northridge, California
  - Riverside, California
  - San Diego, California
  - Wheat Ridge, Colorado
  - New Britian, Connecticut
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - North Miami, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Decatur, Georgia
  - Smyrna, Georgia
  - Boise, Idaho
  - Overland Park, Kansas
  - Rockville, Maryland
  - Boston, Massachusetts
  - Braintree, Massachusetts
  - Brighton, Massachusetts
  - Brockton, Massachusetts
  - Cambridge, Massachusetts
  - Watertown, Massachusetts
  - Farmington Hills, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Clementon, New Jersey
  - Morestown, New Jersey
  - Lawerence, New York
  - New York, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Salem, Oregon
  - Springfield, Oregon
  - Conshohocken, Pennsylvania
  - Emmaus, Pennsylvania
  - Philadelphia, Pennsylvania
  - Scotland, Pennsylvania
  - Anderson, South Carolina
  - Madison, Tennessee
  - Memphis, Tennessee
  - Selmer, Tennessee
  - Austin, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Lakewood, Washington
  - Seatle, Washington
  - Spokane, Washington
  - Madison, Wisconsin

REFERENCES:
- [Result] Snedecor SJ, Botteman MF, Schaefer K, Sarocco P, Barry N, Pickard AS. Economic outcomes of eszopiclone treatment in insomnia and comorbid major depressive disorder. J Ment Health Policy Econ. 2010 Mar;13(1):27-35. PMID 20571180
- [Result] Fava M, Schaefer K, Huang H, Wilson A, Iosifescu DV, Mischoulon D, Wessel TC. A post hoc analysis of the effect of nightly administration of eszopiclone and a selective serotonin reuptake inhibitor in patients with insomnia and anxious depression. J Clin Psychiatry. 2011 Apr;72(4):473-9. doi: 10.4088/JCP.09m05131gry. Epub 2010 Nov 2. PMID 21208574